CLINICAL TRIAL: NCT00753961
Title: EFFECT OF THE CONSUMPTION OF FERMENTED DAIRY DRINK ON COMMON INFECTIONS IN SHIFT-WORKERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NU289
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Shiftworkers; volunteers
MeSH Terms: interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): fermented dairy product
  Interventions: Other: fermented dairy product
- 2 (Placebo Comparator): non fermented acidified dairy product.
  Interventions: Other: non fermented dairy product

INTERVENTIONS:
Other: fermented dairy product — fermented dairy product (2 bottles/day during 16 weeks)
  Arms: 1
Other: non fermented dairy product — non fermented dairy product (2 bottles/day during 16 weeks)
  Arms: 2

SUMMARY:
This clinical study plans to investigate the effect of the consumption of a fermented dairy drink on the occurrence of common infections. This study will be performed in a healthy adult population of shift workers.

ELIGIBILITY:
Inclusion Criteria:

* Male/female subjects aged 18 to 65 years (bounds included)
* Healthy subjects.
* Subjects working in two- or three-shift work including night work

Exclusion Criteria:

* Subject with any food allergy
* Subject in a situation that, in the investigator opinion, could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1340 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of common infectious diseases during the 16 weeks of study product consumption | 0-16 weeks

SECONDARY OUTCOMES:
Mean duration of common infectious diseases during the 16 weeks of study product consumption. | 0-16 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- SGS, Antwerp, Belgium
- Therapharm, Caen, France
- Hospital de la Santa Creu, Barcelona, Spain
- VEEDA, Plymouth, United Kingdom